CLINICAL TRIAL: NCT01109537
Title: Thalamic and Anterior Cingulate Cortex GABA and Glutamate in Restless Legs Syndrome: A 1-HMRS Study
Brief Title: Altered Brain GABA and Glutamate in Restless Legs Syndrome
Acronym: RLS
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, John W. Winkelman, MD, PhD, Associate Professor of Psychiatry, Harvard Medical School, Brigham and Women's Hospital
Other Study IDs: BWH-2010-12345
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome (RLS); GABA; Glutamate; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RLS Diagnosis
- Healthy Controls

SUMMARY:
The purpose of the study is to understand the brain chemistry of people with Restless Legs Syndrome (RLS). The primary hypothesis is that patients with RLS will have reduced GABA levels in their Thalamus and elevated Glutamate levels in their Anterior Cingulate Cortex. The study will use MRS imaging to examine the regional levels of these neurochemicals, GABA and Glutamate, in the brain.

DETAILED DESCRIPTION:
The study will involve a screening visit, a washout period for those taking RLS medications, a night of actigraphy, an overnight polysomnogram, an MRI scan, and an MRS scan. The polysomnography and MR scan visits will occur on consecutive days.

Visit 1: Screening Visit

The informed consent process for the study will be completed and a signed informed consent form will be obtained. All subjects with RLS will undergo a clinical interview in order to confirm or exclude an RLS diagnosis consistent with the International Restless Legs Syndrome Study Group criteria and to determine the presence of any psychiatric or medical disorders. The following study assessments will be completed:

* International Restless Legs Syndrome Scale (IRLS) (RLS subjects only)
* Clinical Global Impression-Severity (CGI) (RLS subjects only)
* Insomnia Severity Index (ISI)
* Beck Depression Inventory
* Pittsburgh Sleep Quality Index (PSQI)
* Hamilton Anxiety Scale (HAM-A)
* Sleep Health Centers Questionnaire
* Metal implant questionnaire

All women will have a urine pregnancy test and all subjects will have a urine sample for drug screening collected.

Washout Period

Subjects in the RLS group will be required to discontinue their RLS medications at least 48 hours prior to the PSG.

Actigraphy

An actigraph will be used to record limb movements of both legs the night before the PSG. The actigraph will be worn from the subjects' bedtime until the subjects' final wake time Subjects will also record their bedtime and wake time on the Actigraphy Data Form. Data from the night of actigraphy will be used to monitor subjects' sleep.

Visit 2: Polysomnography (PSG) The PSG will occur on the night prior to the MRS visit. The time of lights out during all PSG sessions will be determined for each subject based on self report of usual bedtime.

Channels will include an electroencephalograph (EEG), an electro-oculogram (EOG), a submental electromyography (EMG), EMG of both anterior tibialis muscles (separate channels for each leg), oral/nasal airflow, pulse oximetry, and respiratory effort. The PSG will be analyzed for traditional sleep staging. Measures from the PSG will include Sleep Onset Latency (SOL), Wake After Sleep Onset (WASO), Sleep Efficiency (SE), N-REM and REM percentages, Periodic Limb Movement Index (PLMI) and PLMs associated with arousal per hour of sleep (PLMAI).

Visit 3: MR scans

Following visits 1 and 2, qualified subjects will undergo Magnetic Resonance brain scans the Brain Imaging Center of McLean Hospital in Belmont, MA. Prior to MR scanning, subjects will be questioned for a second time about the presence of metallic implants and fragments or any other contraindications to MR imaging. They will be asked about recent alcohol, drug (licit and illicit), and caffeine use. They will also be asked to provide a urine sample for drug screening. Women will take a urine pregnancy test. Also, since brain GABA levels can be affected by the menstrual cycle, women will be scheduled to have their MR scans during the first portion of their menstrual cycle. Subjects will also be asked to complete the following assessments before the MR scans:

* IRLS (modified)
* Medical Outcomes Study Sleep Scale (modified) (MOS)
* Profile of Mood States (POMS)
* Patient Global Impression-Severity (PGI-S)
* State Trait Anxiety Inventory (STAI)

Subjects will undergo proton magnetic resonance spectroscopy (MRS) at 4T. In addition, in accordance with the McLean Hospital Neuroimaging center guidelines, subjects will additionally have a MR screening scan at either 1.5T or 3T. All MR recordings will be obtained using parameters that are within FDA safety guidelines for exposure to static magnetic fields, radio-frequency energy deposition, magnetic field switching rates and acoustic noise levels. GABA and glutamate levels will be derived from MRS Scan at 4T. Subjects will be in each scanner for approximately one hour. At the conclusion of each scan, subjects will be queried regarding any adverse effects related to MR scans. The subject will have completed the study at the conclusion of the MR scans.

During the MRS at 4T, patients will complete a modified Suggested Immobilization Test (SIT). During the SIT, the subjects will be asked by study staff to verbally rate the level of discomfort in their legs on a scale from 1 (no discomfort) to 10 (extreme discomfort). Subjects will be asked to make a rating in five minute intervals over one hour.

In the case that MR scans on the 1.5T/3T and 4T MR scanners cannot be coordinated on the same visit day at the McLean Brain Imaging center due to scheduling conflicts, the subject will be offered the opportunity to return to McLean to have the remaining scan on a separate day. Subjects will still be offered $50 for completion of each scan. Also, in the case that the data collected during MR imaging is not usable (due to technical problems with the scanner, excessive noise in the measurement, etc.), the subject may be contacted and offered a repeat MRS scan on a separate date. Subjects will be compensated an additional $100 for completion of such a repeat MRS scan.

The Primary Endpoints of this protocol are regional GABA and glutamate levels derived from 4T MRS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years of age
* Subjects with a diagnosis of RLS using the International RLS Study Group (IRLSSG) criteria
* Subjects with a history of RLS symptoms at least 15 nights in the prior month, or, if on treatment, this frequency of symptoms before treatment was started

Exclusion Criteria:

* Subjects who are unable to discontinue prohibited medications prior to sleep study and 1H-MRS. These include any CNS-active medications. For RLS subjects, RLS-related medications (e.g. dopaminergic agents and alpha 2-delta agents) must be discontinued a minimum of 48 hours prior to PSG. In the RLS group, benzodiazepines must be discontinued a minimum of one week prior to PSG. For normal controls with regular treatment (>1 time/wk) with CNS active agents within 1 month of screening visit will also be excluded.
* Subjects with an active or unstable major psychiatric disorder requiring further treatment (e.g., major depressive disorder). Subjects with clinically significant depression, or with clinically significant anxiety, or who, in the investigator's judgment might require intervention with either pharmacological or non-pharmacological therapy over the course of the study.
* Subjects with clinical evidence of any untreated moderate to severe sleep disorder other than RLS (forRLS group) (e.g. obstructive sleep apnea, insomnia, narcolepsy, delayed sleep phase syndrome, etc.) within the preceding year
* Subjects with an apnea-hypopnea index (AHI) > 15 at the polysomnography visit
* Subjects who consume beverages containing more than 400mg of caffeine per day
* Subjects who consume more than 14 alcoholic units in any week, or more than 5 alcoholic units in any single day, over the month preceding the screening visit.
* Females who are pregnant or lactating
* Subjects with a history of neurologic illness (e.g. brain neoplasm, multiple sclerosis), significant or unstable medical illness (e.g. congestive heart failure, diabetes mellitus), or history of significant head trauma or loss of consciousness > 30 minutes
* Subjects who have positive urine drug screening (phencyclidine, cocaine, amphetamines, tetrahydrocannabinol, and opiates) at the screening visit or at the MRS visit.
* Contraindications to MRS scans, including:
* Cardiac pacemakers
* Aneurysm clips and other vascular stents, filters, clips or other devices
* Prosthetic heart values
* Other prostheses
* Neuro-stimulator devices
* Implanted infusion pumps
* Cochlear (ear) implants
* Ocular (eye) implants or known metal fragments in eyes
* Exposure to shrapnel or metal filings (sheetmetal workers, welders, and others)
* Other metallic surgical hardware in vital areas
* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female subjects who have RLS or are normal controls will be recruited from the greater Boston metropolitan area. We anticipate enrolling 70 subjects with RLS and 70 normal controls, under a plan to complete 15 subjects in each group.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2010-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Regional GABA and glutamate levels derived from 4T MRS. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John W Winkelman, MD, PhD, Principal Investigator — Sleep Health Centers, Brigham and Women's Hospital
Locations (1):
- Sleep HealthCenters, Brighton, Massachusetts, United States

REFERENCES:
- [Background] Bucher SF, Seelos KC, Oertel WH, Reiser M, Trenkwalder C. Cerebral generators involved in the pathogenesis of the restless legs syndrome. Ann Neurol. 1997 May;41(5):639-45. doi: 10.1002/ana.410410513. PMID 9153526
- [Background] Price DD. Psychological and neural mechanisms of the affective dimension of pain. Science. 2000 Jun 9;288(5472):1769-72. doi: 10.1126/science.288.5472.1769. PMID 10846154
- [Background] Cervenka S, Palhagen SE, Comley RA, Panagiotidis G, Cselenyi Z, Matthews JC, Lai RY, Halldin C, Farde L. Support for dopaminergic hypoactivity in restless legs syndrome: a PET study on D2-receptor binding. Brain. 2006 Aug;129(Pt 8):2017-28. doi: 10.1093/brain/awl163. Epub 2006 Jul 1. PMID 16816393
- [Background] von Spiczak S, Whone AL, Hammers A, Asselin MC, Turkheimer F, Tings T, Happe S, Paulus W, Trenkwalder C, Brooks DJ. The role of opioids in restless legs syndrome: an [11C]diprenorphine PET study. Brain. 2005 Apr;128(Pt 4):906-17. doi: 10.1093/brain/awh441. Epub 2005 Feb 23. PMID 15728657
- [Background] Spiegelhalder K, Feige B, Paul D, Riemann D, van Elst LT, Seifritz E, Hennig J, Hornyak M. Cerebral correlates of muscle tone fluctuations in restless legs syndrome: a pilot study with combined functional magnetic resonance imaging and anterior tibial muscle electromyography. Sleep Med. 2008 Jan;9(2):177-83. doi: 10.1016/j.sleep.2007.03.021. Epub 2007 Jul 16. PMID 17638594
- [Background] Etgen T, Draganski B, Ilg C, Schroder M, Geisler P, Hajak G, Eisensehr I, Sander D, May A. Bilateral thalamic gray matter changes in patients with restless legs syndrome. Neuroimage. 2005 Feb 15;24(4):1242-7. doi: 10.1016/j.neuroimage.2004.10.021. Epub 2004 Dec 8. PMID 15670702
- [Background] Winkelman JW, Redline S, Baldwin CM, Resnick HE, Newman AB, Gottlieb DJ. Polysomnographic and health-related quality of life correlates of restless legs syndrome in the Sleep Heart Health Study. Sleep. 2009 Jun;32(6):772-8. doi: 10.1093/sleep/32.6.772. PMID 19544754
- [Background] Kushida CA, Allen RP, Atkinson MJ. Modeling the causal relationships between symptoms associated with restless legs syndrome and the patient-reported impact of RLS. Sleep Med. 2004 Sep;5(5):485-8. doi: 10.1016/j.sleep.2004.04.004. PMID 15341894